CLINICAL TRIAL: NCT06112262
Title: Comparison of the Effecta and Drawbacks of Heparin Versus Hirudin Drugs in Haemodialysis Patients in Assiut University Hospitals
Brief Title: Comparison Between Haparin and Herodin in HD
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Basma Rabiey (Other)
Responsible Party: Sponsor-Investigator, Basma Rabiey, Principal investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: heparin and herodin in HD
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Haemodialysis
MeSH Terms: interventions — Heparin; Hirudins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heparin and Hirudin (Experimental): Anticoagulant in Hemodialysis
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Heparin — Comparison between heparin and hirudin
  Other Names: Hirudin

SUMMARY:
The goal of this study is to compare the efficacy and drawbacks of Heparin and Hirudin in Haemodialysis patients. The main question it aims to answer is:

which drug is more safe in Haemodialysis?

DETAILED DESCRIPTION:
Extracorporeal thrombogenesis is a major problem associated with haemodialysis. The composition of the artificial membrane in the extracorporial system and large surface area to which the blood is exposed, contribute significantly to activation of the coagulation cascade and platelets. The use of anticoagulant is to prevent thrombotic occlusion of the dializer to ensure effective dialysis.

The most common anticoagulant options for Hemodialysis include unfractionated heparin (UFH), low-molecular weight heparin (LMWH), thrombin antagonists, and platelet inhibiting agents. The choice of anticoagulant for Haemodialysis should be determined by patient characteristics, local expertise, and ease of monitoring.

Heparins are currently the anticoagulants of choice in long-term haemodialysis (HD), but because of their shortcomings, including the increasing incidence of heparin-induced thrombocytopenia (HIT II), alternative anticoagulation is necessary, as there are several complication associated with its long term use, They include thrombocytopenia, increase bleeding tendency, osteoporosis, increase lipolytic activity and change of lipid pattern, activation of of lipolysis also leads to immunosuppressive effect.

Hirudin the most potent natural inhibitor of thrombin, it is a direct thrombin inhibitor and does not require endogenous cofactors. Hirudin inhibits all actions of thrombin and so effectively inhibit coagulation and prevent heparin resistant arterial type thrombosis when given in large enough doses. Hirudin has no adverse effect when it is used into human, because it is pharmacologically inert. Hirudin is also a weak immunogen.

Few researches evaluate the efficacy and drawbacks of Hirudin in HD patients.

ELIGIBILITY:
Inclusion Criteria:

1. patient age between 18:70
2. Haemodialysis duration less than 6 months
3. Agree to participate in the study

Exclusion Criteria:

1. AKI
2. patients with impaired coagulation profile
3. Decompensated liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of bleeding events and efficacy of dialysis during dialysis | Baseline
  patients will be investigated with aPTT before and after each of the following sessions (HD1, HD4, HD8), CBC/ week, number of clotting events, number of bleeding tendency, duration of fistula closure, to assess anticoagulant efficacy , and BUN, Serum creatinine, urea reduction ratio to assess dialysis efficacy.

REFERENCES:
- [Background] Dangas GD, Lefevre T, Kupatt C, Tchetche D, Schafer U, Dumonteil N, Webb JG, Colombo A, Windecker S, Ten Berg JM, Hildick-Smith D, Mehran R, Boekstegers P, Linke A, Tron C, Van Belle E, Asgar AW, Fach A, Jeger R, Sardella G, Hink HU, Husser O, Grube E, Deliargyris EN, Lechthaler I, Bernstein D, Wijngaard P, Anthopoulos P, Hengstenberg C; BRAVO-3 Investigators. Bivalirudin Versus Heparin Anticoagulation in Transcatheter Aortic Valve Replacement: The Randomized BRAVO-3 Trial. J Am Coll Cardiol. 2015 Dec 29;66(25):2860-2868. doi: 10.1016/j.jacc.2015.10.003. Epub 2015 Oct 15. PMID 26477635